CLINICAL TRIAL: NCT01042821
Title: Treatment of Anal Fistulas by Partial Rectal Wall Advancement Flap or Mucosal Advancement Flap: a Prospective Randomized Study
Brief Title: Treatment of Anal Fistulas Advancement Flap
Acronym: flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: dr waeil khafagy, Mansoura university hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anal fistula
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2005-05

CONDITIONS: Anal Fistula
Keywords: anal fistula; advancement flap; incontinence
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- partial rectal wall advancement flap (Active Comparator): The flap comprised mucosa, submucosa and circular muscle fibers. It is raised from the dentate line and mobilized 4-6 cm cephaled and advanced to the new dendentate line (1 cm below the dentate line) and sutured with absorbable sutures (vicryl; ethicone 3/0). Also the defect is closed with absorbable sutures.
  Interventions: Procedure: partial rectal wall advancement flap
- Group 2 (Active Comparator): The flap comprised mucosa, submucosa only
  Interventions: Procedure: mucosal advancement flap

INTERVENTIONS:
Procedure: partial rectal wall advancement flap — The flap comprised mucosa, submucosa and circular muscle fibers. It is raised from the dentate line and mobilized 4-6 cm cephaled and advanced to the new dendentate line (1 cm below the dentate line) and sutured with absorbable sutures (vicryl; ethicone 3/0). Also the defect is closed with absorbable sutures.
  Other Names: Group 1
  Arms: partial rectal wall advancement flap
Procedure: mucosal advancement flap — Fistulectomy, closure of internal sphincter and rectal advancement flap includes mucosa and submucosal layer sutured 1cm below the level of internal opening
  Other Names: advancement flap
  Arms: Group 2

SUMMARY:
This study comprises a prospective study of 40 patients with transphincteric anal fistula. The patients were classified into two groups: Group I: Fistulectomy, closure of internal sphincter and rectal advancement flap includes mucosa, submucosa, and circular muscle layer sutured 1cm below the level of internal opening. Group II: The same as group one but the flap includes only mucosa and submucosa.

DETAILED DESCRIPTION:
This study comprises a prospective study of 40 patients with transphincteric anal fistula. They were referred to our colorectal surgery unit, Mansoura University Hospital during the period from May 2005 to May 2008. Patients with acute sepsis, specific cause of fistula, strictured anorectum, and any degree of incontinence were excluded from the study.

All patient were evaluated by digital examination, procto-sigmoidoscopy, fistulography and MRI fistulography without contrast media, using a 1.5 Tesla super conducting magnet (Magnetom Symphony MRease VA12 Siemens medical system), (either STIR or SPIR in addition to T1 weighted or T2 weighted sequences). Axial, coronal and sometimes sagittal planes were used. Preoperative assessment of anal sphincter dysfunction was done by conventional manometry using a standard low compliance water perfusions system and eight-channels catheters with pressure transducer connected to 5.5 mm manometric probe with spirally located ports at 0.5cm interval, which measured along the length of the anal canal, as well as inflatable rectal balloon. The protocol of performance is stationary pull through technique with recording the functional length of the anal canal (FL), mean maximum resting pressure in the anal canal (MRP), mean maximum squeeze pressure in the anal canal (MSP). Pressure was recorded using a computerized recording device (MMS ;Holland) which included menu-driven software to aid with data acquisition. Data were analyzed with the use of a complied software package that automatically produced numeric reports and graphs.

The patients were then classified into 2 groups. After carefully explaining the purpose of the study, an informed consent was taken from every patient. Group I: Fistulectomy, closure of internal sphincter with loose vicryl 3(0) suture and rectal advancement flap (the length 5cm of the flap is twice its width) includes mucosa, submucosa, circular muscle layer sutured 1cm below the level of internal opening. Group II: The same as group one but the flap includes only mucosa and submucosa.

Surgical technique:

Fleet enema was used for preoperative bowel preparation in all cases. Operation was done under general anesthesia in the lithotomy position. Prophylactic antibiotics were used with ciprofloxacin 500 mg and metronidazole 500 mg preoperatively and twice daily for 5 days. Examination under anaesthesia (EUA) was firstly performed and the extent of the disease was established by cannulating the fistulas with probes and by laying open all primary tracts, extensions, and abscesses. All the incisions and dissections were made by electrocautery. The standard procedure was to perform core fistulectomy and traversing the external sphincter until the internal sphincter was exposed the track was then transected. The crypt-bearing tissue around the internal opening of the fistula is excised, if there is difficulty in excising the main tract, the granulation tissue of the remaining tract is scraped with a curette. Advancement flap was constructed in both group.

1. Group I: - The flap comprised mucosa, submucosa and circular muscle fibers. It is raised from the dentate line and mobilized 4-6 cm cephaled and advanced to the new dendentate line (1 cm below the dentate line) and sutured with absorbable sutures (vicryl; ethicone 3/0). Also the defect is closed with absorbable sutures.
2. Group II: - The flap comprised mucosa, submucosa only.

Rectal pack was removed after 24 hours. The patients were allowed to drink freely for 5 days, then normal diet and laxatives. The external fistulectomy wound was dressed daily. Histopatho;ogical examination of all excised fistulous tract was done.

1. Follow up of our patients had been done for about 12 months with clinical assessment of the patients as regard. Incidence of any postoperative complications as bleeding, haematoma, ecchymosis, and disruption. Incidence of any degree of postoperative incontinence according to Cliveland clinic incontinence Score (Rockwood et al., 1999). Recurrence was defined as a discharge or abscess arising in the same area or by obvious evidence of fistulation.

Postoperative assessment of physioanatomical changes in the anal sphincter using anal manometry: 6 months post-operative after wound healing to measure MRP & MSP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transphincteric anal fistula

Exclusion Criteria:

* Patients with acute sepsis, specific cause of fistula, strictured anorectum, and any degree of incontinence

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
RECURRENCE OF THE FISTULA | 12 months

SECONDARY OUTCOMES:
healing, complication, patient satisfaction | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Wael Khafagy, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

REFERENCES:
- [Result] Ortiz H, Marzo J, Ciga MA, Oteiza F, Armendariz P, de Miguel M. Randomized clinical trial of anal fistula plug versus endorectal advancement flap for the treatment of high cryptoglandular fistula in ano. Br J Surg. 2009 Jun;96(6):608-12. doi: 10.1002/bjs.6613. PMID 19402190
- [Result] Dixon M, Root J, Grant S, Stamos MJ. Endorectal flap advancement repair is an effective treatment for selected patients with anorectal fistulas. Am Surg. 2004 Oct;70(10):925-7. PMID 15529853
- [Result] Christoforidis D, Pieh MC, Madoff RD, Mellgren AF. Treatment of transsphincteric anal fistulas by endorectal advancement flap or collagen fistula plug: a comparative study. Dis Colon Rectum. 2009 Jan;52(1):18-22. doi: 10.1007/DCR.0b013e31819756ac. PMID 19273951
- [Result] Chung W, Kazemi P, Ko D, Sun C, Brown CJ, Raval M, Phang T. Anal fistula plug and fibrin glue versus conventional treatment in repair of complex anal fistulas. Am J Surg. 2009 May;197(5):604-8. doi: 10.1016/j.amjsurg.2008.12.013. PMID 19393353
- [Result] Dubsky PC, Stift A, Friedl J, Teleky B, Herbst F. Endorectal advancement flaps in the treatment of high anal fistula of cryptoglandular origin: full-thickness vs. mucosal-rectum flaps. Dis Colon Rectum. 2008 Jun;51(6):852-7. doi: 10.1007/s10350-008-9242-3. Epub 2008 Mar 4. PMID 18317841
- See also: Mansoura university hospital — http://www.mans.eun.eg/